CLINICAL TRIAL: NCT00782392
Title: Bioavailability and Dosing of an Oral Monosaccharide Supplement in Adults and Effects on Resting Brain Activity
Brief Title: Bioavailability and Dosing of a Monosaccharide Supplement in Adults
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: University of Arkansas (Other); United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Joanne S. Szabo, M.D., University of Arkansas for Medical Sciences
Other Study IDs: 45092
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2011-05

CONDITIONS: Healthy Males
Keywords: Nutrition; Infant Formula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
We are developing an oral supplement of carbohydrates to be added to infant formulas in order to improve brain development, immune function, and overall health of infants and children. After a careful review of what is known about these sugars, there is very little information regarding their use in infants and children, although there is some information in adults and animals.

Many of these sugars have been used in a glyco-nutritional supplement in adults and children, with minimal or no reported side effects.

We are developing a custom blend of important individual sugars, and need information regarding their dosing and blood concentrations following oral intake of the carbohydrate supplement. Timed blood samples following the carbohydrate supplement will provide us with a better understanding of the most effective dose and the metabolism of these sugars in adults. This will give us the preliminary information we need for developing an oral supplement of special sugars that can be added to infant formulas to help improve brain development and immune function in infants and children.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian (non-hispanic)
* Male
* Age 18-28
* Regularly eat breakfast
* Healthy
* BMI within normal limits (18.5 - 24.9)
* English speaking

Exclusion Criteria:

* History of smoking, more than occasional alcohol use, or drug use.
* Chronic medical diagnosis
* Medications that may interfere with the study

Ages: 18 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Caucasian Males
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2007-01; Primary Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States